CLINICAL TRIAL: NCT00007748
Title: CSP#470 - A Randomized, Multi-Center, Controlled Trial of Multi-Modal Therapy in Veterans With Gulf War Illnesses
Brief Title: Exercise and Behavioral Therapy Trial (EBT).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 470
Record Dates: First submitted 2000-12-29; First posted 2001-01-01 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Persian Gulf Syndrome
Keywords: aerobic exercise; cognitive behavioral therapy; CBT; Gulf War Illnesses; GWI
MeSH Terms: conditions — Persian Gulf Syndrome | interventions — Exercise; Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Aerobic exercise
Behavioral: Cognitive behavioral therapy

SUMMARY:
This trial is a study of Gulf War era veterans who have unexplained chronic medical symptoms such as pain, fatigue, and/or cognitive difficulties. The treatments to be studied, cognitive behavior therapy (CBT) and aerobic exercise, have been shown to be effective in alleviating symptoms in individuals with other similar types of illnesses, such as chronic fatigue syndrome and fibromyalgia. This is a Phase 3, 2X2 factorial designed study. All study participants are assigned to one of four treatment groups - CBT and aerobic exercise, aerobic exercise alone, CBT alone or usual and customary care. This study durations is 28 months; 1092 participants were enrolled and will be followed in clinic at 3, 6 and 12 months after enrollment.

DETAILED DESCRIPTION:
Primary Hypothesis:

The primary hypothesis is that both aerobic exercise and cognitive behavioral therapy (CBT) will significantly improve physical function (as measured by the Physical Component Summary Scale of the SF-36V) in veterans with Gulf War Veterans' Illnesses (GWVI), and the combination of cognitive behavioral therapy and aerobic exercise will be more beneficial than either therapy alone.

Secondary Hypotheses:

1. Both aerobic exercise and CBT will lead to improvements in the cardinal symptoms of GWVI: pain, fatigue and cognitive difficulties.
2. Both aerobic exercise and CBT will lead to decreased levels of distress in persons with GWVI.
3. Both aerobic exercise and CBT will lead to improvements in emotional functioning in persons with GWVI.

Primary Outcomes: Improvement on the Physical Component Summary Scale of the SF-36V of more than 7 units at one year relative to baseline.

Interventions: Twelve one-hour weekly sessions of Cognitive behavioral therapy, aerobic exercise, the combination of the two therapies (12 one-hour sessions of CBT and 12 one-hour sessions of aerobic exercise) and a control group that receives usual and customary care.

Study Abstract: This trial was a study of Gulf War era veterans who have unexplained chronic medical symptoms such as pain, fatigue, and/or cognitive difficulties. All Gulf War veterans who were deployed to the South West Asia theater of operations between August 1990 and August 1991 were eligible for the study if they had at least two of the following three symptoms that began after August of 1990, lasting for more than six months and occurring up to present: 1. fatigue that limits usual activities (work, recreation, or social), 2. musculoskeletal pain involving two or more regions of the body, and neuro-cognitive dysfunction (self-reported difficulties in memory, concentration, or attention). Veterans who met enrollment criteria were randomized to one of four treatment arms: 1. CBT plus aerobic exercise, 2. aerobic exercise alone, 3. CBT alone, and 4. usual and customary care. Treatment was given for three months in group format. The CBT and exercise groups met for one hour, once a week for 12 weeks for a total of 12 hourly sessions. The interventions were standardized and all investigators were trained in the use of these methods prior to start up of the trial. The target sample size was 1064 veterans with GWVI to be accrued from 20 Medical Centers (18 VA and 2 DOD). All veterans were followed for one year and outcomes measured at 3 months (immediately following the end of treatment), 6 months and 12 months after enrollment.

The study was kicked-off in April 1999 and enrollment ended on September 5, 2000, during which 1092 veterans were randomized. Patient follow-up concluded on September 30, 2001 and the final DSMB meeting was held on November 28, 2001. The major finding was that there were no significant differences in the proportion of veterans who reported an improvement in physical function at one year among the treatment groups (11.5% for usual care, 11.7% for exercise, 18.4% for CBT and 18.5% for CBT + exercise). However, statistically significant improvements in fatigue, cognitive symptoms, distress, and mental health functioning were observed with exercise alone and with exercise plus CBT compared to usual care. CBT alone had a statistically significant effect on cognitive symptoms and in mental health functioning. Except for affective pain, which improved with CBT alone or with exercise, neither treatment had a significant effect on the other three measures of pain. In summary, neither exercise nor CBT had a significant impact on physical function for veterans with GWVI but both treatments, especially exercise, resulted in improvement in fatigue, cognitive symptoms, distress and mental health functioning.

Results embargoed until publication.

ELIGIBILITY:
Gulf War era veterans deployed to the South West Asia theater of operations between August 1990 and August 1991 who have two of the following three symptoms that began after 1990 lasting more than 6 months and continuing to present - fatigue that limits usual activities (work, recreation or social), musculoskeletal pain involving more than one region of the body or neurocognitive dysfunction (self-reported difficulties in memory, concentration, or attention).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1064
Dates: Start 1999-03; Study Completion 2001-08

CONTACTS AND LOCATIONS:
Locations (25):
- United States (24):
  - Birmingham Vamc Birmingham Vamc, Birmingham, Alabama
  - Birmingham Vamc, Birmingham, Alabama
  - Naval Health Research Center, San Diego, San Diego, California
  - San Francisco Vamc, San Francisco, California
  - VA CT Healthcare System, West Haven, West Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Uniformed Services University, Bethesda, Maryland
  - Boston Vamc, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - John Cochran VAMC, Saint Louis, St Louis, Missouri
  - VA New Jersey Health Care System, East Orange, East Orange, New Jersey
  - Vamc - Albuquerque, Albuquerque, New Mexico
  - New York Harbor VA Healthcare System, Brooklyn Campus, Brooklyn, New York
  - Fargo Vamc, Fargo, North Dakota
  - Vamc - Dayton, Dayton, Ohio
  - Portland Vamc, Portland, Oregon
  - Philadelphia Vamc, Philadelphia, Pennsylvania
  - Houston Vamc, Houston, Texas
  - Audie L. Murphy Memorial Veterans Hospital, San Antonio, San Antonio, Texas
  - White River Junction Vamc, Burlington, Vermont
  - White River Junction Vamc, White River Jct., Vermont
  - Richmond Vamc, Richmond, Virginia
  - VA Puget Sound Healthcare System, Seattle Division, Seattle, Washington
- San Juan Vamc, San Juan, Puerto Rico